CLINICAL TRIAL: NCT04896164
Title: Phase III Randomized, Double Blind, Placebo Controlled Study of Curcumin to Reduce Mucositis in Autologous Transplant Setting
Brief Title: Randomized Trial of Curcumin to Reduce Mucositis in Autologous Transplant Setting
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Navin Khattry, Professor and BMT convener, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 900503; CTRI/2018/09/015846 (Registry Identifier: Clinical Trials Registry - India (CTRI))
Record Dates: First submitted 2021-05-15; First posted 2021-05-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Oral Mucositis (Ulcerative)
Keywords: Curcumin; Mucositis; Autologous stem cell transplant
MeSH Terms: conditions — Stomatitis; Ulcer; Mucositis

STUDY DESIGN:
Intervention Model Description: Patients receiving high dose chemotherapy with any of the conditioning regimens specified in the inclusion criteria will be randomized in two arms. Central telephonic randomization will be carried out with the help of a computer generated random sequence using permuted blocks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The test drug and the placebo are available in USP grade plastic bottles. The bottles are identical in all respect. Each bottle have a unique identifier number provided by the manufacturer. The transplant physician, patients and the blinded statistician will remain blinded to the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational arm (Experimental): Patients in the investigational arm will receive curcumin lozenges (4 gm BD containing 400 mg curcumin BD) as prophylaxis from two days prior to receiving high dose chemotherapy .
  Interventions: Drug: Curcumin Lozenges
- Control arm (Placebo Comparator): patients in the control arm will receive matching placebo lozenges from two days prior to receiving high dose chemotherapy
  Interventions: Other: Placebo Lozenges

INTERVENTIONS:
Drug: Curcumin Lozenges — Curcumin lozenges (each containing 100 mg of curcumin) will be given at a dose of 4 lozenges (total dose 400 mg curcumin) BD. Formulation is Solid Lipid Curcumin Particle (SLCP). Oral curcumin lozenges will be given from two days prior to receiving high dose chemotherapy till day+28 of transplant.
  Other Names: Longvida (Pharmanza Herbal Pvt Ltd.)
  Arms: Investigational arm
Other: Placebo Lozenges — Placebo lozenges will be given from two days prior to receiving high dose chemotherapy till day+28 of transplant.
  Arms: Control arm

SUMMARY:
Mucositis is a very common complication in bone marrow transplant setting. It is a result of injury to the gut caused by high dose chemotherapy. Currently there are no universal protocols that have been accepted as a standard to prevent and treat mucositis in the transplant setting. Post transplant upto 80% of patients suffer from a severe mucositis. Proinflammatory cytokines play a major role in the development of mucositis. Interventions that decrease the levels of these cytokines may be beneficial in preventing mucositis. This study is aimed at evaluating the role of curcumin in reducing cytokine levels and the incidence and duration of mucositis in patients undergoing autologous stem cell transplantation.

DETAILED DESCRIPTION:
Mucositis is an inevitable side-effect of intensive conditioning therapy used for hematopoietic stem cell transplantation and affects the quality of life of patients undergoing transplant. The incidence of oral mucositis (WHO grades 3/4 ) with certain myeloablative conditioning regimens has been reported in up to 90% with range of severe mucositis (WHO grade 3/4) from 10 to 78%. Pro-inflammatory cytokines such as IL-1, IL-6, IL-8, IL-17, TNF-α, TGF-B, IFN-γ and certain prostaglandins play a central role in its pathogenesis. Transcription factors such as NF-kappa B, modify the genetic expression of these cytokines and enzymes which are critical in producing tissue damage.

A number of agents and methods have been investigated to prevent or reduce mucositis in transplant setting. Some of them are amifostine, caphasol, palifermin, cryotherapy, chlorhexidine, glutamine, GM-CSF, histamine, misoprostol, laser therapy and traumeel, but only palifermin and cryotherapy have shown significant benefit.

Curcumin, polyphenol derivative with low toxicity profile, is commonly used in India for its anti-inflammatory actions. Curcumin inhibits various inflammatory cytokines through inhibition of Nuclear Factor Kappa- β. It is derived from the plant Curcuma longa. In vitro studies have shown potent anti-inflammatory activity at concentrations of 1 umol/L.

The investigators conducted the first study evaluating the role of curcumin on oral mucositis in transplant setting. In this pilot study (n=40), patients who received curcumin lozenges (n=30) had decreased levels of salivary TGF-β, IL-17 and serum PGE2 compared to patients who did not receive the curcumin lozenges (n=10). Patients who received the curcumin lozenges had higher levels of serum IL-8 which is a prohealing cytokine. The incidence of grade 3 and 4 oral mucositis and diarrhea was less in those who received curcumin lozenges. Curcumin lozenges were also well tolerated and none of the 30 patients who were administered curcumin developed any treatment related grade 3/4 toxicity. This encouraging data is the basis of the current phase III randomized study comparing curcumin lozenges to placebo, to assess the ability of curcumin to reduce the incidence and duration of oral mucositis in patients undergoing autologous bone marrow transplantation.

The formulation being used is a Solip Lipid Curcumin microParticle (SLCP). The formulation is developed by Pharmanza Herbals Pvt. Ltd., Gujarat, India. Gota et al reported a phase I clinical trial of SLCP where upto 4 grams of the formulation containing 20-30% curcumin was evaluated for safety and pharmacokinetics in patients with high-risk osteosarcoma (Ref). The SLCP formulation showed oral bioavailability of curcumin with linear pharmacokinetics. Average peak plasma concentration of 41 ng/mL was observed at the highest dose level of 4g. All doses were well tolerated and no adverse events were observed. Based on these observations (on safety and bioavailability), and the reported anti-inflammatory properties of curcumin, it was envisaged that it could be potentially useful for the prophylaxis and treatment of oral mucositis following high-dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years and above.
2. Patients who give written informed consent
3. Patients with performance status - 0,1 or 2 (ECOG scale)
4. Patients receiving any of the following high dose chemotherapy regimens for autologous transplant in any indicated malignant disease.

   1. Melphalan- 200 mg/m2 or more (MEL-200 mg/m2)
   2. Busulfan and Melphalan (BuMEL)
   3. Carmustine (BCNU), Etoposide, Cytosine Arabinoside and Melphalan ( BEAM)
5. Patients who have creatinine clearance > 50 ml/min
6. Patients with serum bilirubin levels < 2mg/dl. and serum liver enzymes (ALT or AST or both) lesser than 5 times the upper limit of normal value.

Exclusion Criteria:

1. Patients who are on NSAIDs, aspirin, antioxidants or systemic steroids for more than 3 months and the last dose taken within the last one week.
2. Patients being treated for active infection at the time of starting high dose chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2018-12-16 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 and 4 oral mucositis | Day+28
  In both groups, patients will be evaluated clinically for oral mucositis. The incidence of grade III/IV oral mucositis will be recorded as per WHO grading criteria.

SECONDARY OUTCOMES:
Incidence of any grade of oral mucositis. | Day+28
  In both groups, patients will be evaluated clinically for oral mucositis and grade will be recorded as per WHO grading criteria.
Duration of grade 3 and 4 oral mucositis in both groups | Day+28
  In both groups, duration of oral mucositis will be recorded.
Incidence of use of Total Parenteral Nutrition | Day+28
  Incidence of use of Total Parenteral Nutrition in both groups.
Duration of use of Total Parenteral Nutrition | Day+28
  The duration of use of total parenteral nutrition will be recorded in both groups.
Serum TNF alpha AUC (0-14) | Day+14
  This will be calculated using serum TNF alpha levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary TNF alpha AUC (0-14) | Day+14
  This will be calculated using Salivary TNF alpha levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum Interleukin 1 AUC (0-14) | Day+14
  This will be calculated using Serum Interleukin 1 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary Interleukin 1 AUC (0-14) | Day+14
  This will be calculated using Salivary Interleukin 1 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum Interleukin 6 AUC (0-14) | Day+14
  This will be calculated using Serum Interleukin 6 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary Interleukin 6 AUC (0-14) | Day+14
  This will be calculated using Salivary Interleukin 6 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum Interleukin 8 AUC (0-14) | Day+14
  This will be calculated using Serum Interleukin 8 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary Interleukin 8 AUC (0-14) | Day+14
  This will be calculated using Salivary Interleukin 8 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum Interleukin 17 AUC (0-14) | Day+14
  This will be calculated using Serum Interleukin 17 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary Interleukin 17 AUC (0-14) | Day+14
  This will be calculated using Salivary Interleukin 17 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum TGF-beta AUC (0-14) | Day+14
  This will be calculated using Serum TGF-beta levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary TGF-beta AUC (0-14) | Day+14
  This will be calculated using Salivary TGF-beta levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum Interferon gamma AUC (0-14) | Day+14
  This will be calculated using Serum Interferon gamma levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary Interferon gamma AUC (0-14) | Day+14
  This will be calculated using Salivary Interferon gamma levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Serum Prostaglandin E2 AUC (0-14) | Day+14
  This will be calculated using Serum Prostaglandin E2 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Salivary Prostaglandin E2 AUC (0-14) | Day+14
  This will be calculated using Salivary Prostaglandin E2 levels measured at baseline, day 0, then Monday, Wednesday and Friday till day +14. Using these values, AUC (0-14) will be calculated using linear trapezoidal model.
Plasma curcumin AUC (0-12 hr) | Up to 12 hours from 1st dose
  This will be done using plasma curcumin levels measured within 1 hr of dosing, 0.5-3 hr, 4-6 hr, and 8 - 12 hr post dose on day 7 of starting curcumin or placebo.
Plasma Bis-demethoxycurcumin AUC (0-12 hr) | Up to 12 hours from 1st dose
  This will be done using plasma Bis-demethoxycurcumin levels measured within 1 hr of dosing, 0.5-3 hr, 4-6 hr, and 8 - 12 hr post dose on day 7 of starting curcumin or placebo.
Plasma demethoxycurcumin AUC (0-12 hr) | Up to 12 hours from 1st dose
  This will be done using plasma demethoxycurcumin levels measured within 1 hr of dosing, 0.5-3 hr, 4-6 hr, and 8 - 12 hr post dose on day 7 of starting curcumin or placebo.
Duration of use of analgesics for pain due to oral mucositis | Day+28
  Duration of use of analgesics for pain due to oral mucositis in both groups will be recorded.The severity of pain will be measured using the visual analog pain scale.
Incidence of grade 3 and 4 nausea | Day+28
  In both groups, grade of nausea will be recorded as per CTCAE v 4.0 grading criteria.
Incidence of grade 3 and 4 vomiting | Day+28
  In both groups, grade of vomiting will be recorded as per CTCAE v 4.0 grading criteria.
Incidence of grade 3 and 4 diarrhea | Day+28
  In both groups, grade of diarrhea will be recorded as per CTCAE v 4.0 grading criteria.
Duration of hospital stay | From date of hospital admission until date of hospital discharge assessed up to day +28
  The duration of hospital stay will be recorded in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Navin Khattry, MD, DM, Principal Investigator — Tata Memorial Centre Advanced Centre for Treatment, Research and Education in Cancer
Locations (1):
- Tata Memorial Centre, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No